CLINICAL TRIAL: NCT06727890
Title: The Efficacy and Safety of Compound Danshen Dripping Pill in Patients With Diabetic Microvascular Angina
Brief Title: Compound Danshen Dripping Pill for Diabetic Microvascular Angina
Acronym: MVA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Pan-Pan Hao, Dr., Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDDP for CMVD
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Microvascular Angina
MeSH Terms: interventions — danshen dripping pill

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compound Danshen Dripping Pill (Experimental)
  Interventions: Drug: Danshen Dripping Pill
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Danshen Dripping Pill — Danshen Dripping Pill, 10 pills once, three times a day
  Arms: Compound Danshen Dripping Pill
Drug: Placebo — Placebo, 10 pills once, three times a day
  Arms: Placebo

SUMMARY:
To investigate the efficacy and safety of Compound Danshen Dripping Pill in patients with diabetic microvascular angina pectoris. Long-term follow-up of 1 year will be performed to evaluate the effect of Compound Danshen Dripping Pill on coronary flow reserve and adverse cardiovascular events in patients with coronary microvascular disease.

ELIGIBILITY:
Inclusion Criteria:

History of type 2 diabetes ≧5 years; Repeated chest pain attacks with typical exertional angina pectoris or resting angina pectoris attacks; Coronary normal or stenosis <50%; Ischemic depression in ST segment during resting or exercise; Coronary flow reserve (CFR) of the anterior descending coronary artery < 2.0, or CFR ≧2.0 but acetylcholine activation test is positive; Subjects or their guardians agreed to participate in this study.

Exclusion Criteria:

Previous myocardial infarction or PCI or CABG treatment; Severe arrhythmia; Refractory hypertension or hypertension accompanied by left ventricular wall thickness > 12 mm; Familial hypercholesterolemia; Takayasu arteritis, Kawasaki disease or coronary artery malformation; Pregnant or nursing, or having the intention to give birth within one year; Hepatic or renal dysfunction; Allergic to contrast agents or traditional Chinese medicines; Patients who participated in clinical research of other drugs within 3 months before being selected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of coronary flow reserve measured by three-dimensional echocardiography from baseline to 12 months after follow-up | From baseline to the end of 12-month treatment

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University/Shandong Province Qianfoshan Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Undecided
It might damage the privacy of patients.